CLINICAL TRIAL: NCT01687114
Title: Urinary Proanthocyanidin (PAC) A2 as a Biomarker of Compliance to Intake of Cranberry Products - A Pilot Study
Brief Title: Urinary Proanthocyanidin-A2 as a Biomarker of Compliance to Intake of Cranberry Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Oliver Chen, Research Scientist II, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HNRC2785
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Tract Infection
Keywords: compliance, proanthocyanidin, phenoic acids, cranberry
MeSH Terms: conditions — Urinary Tract Infections; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cranberry juice (Experimental): 27% cranberry juice
  Interventions: Other: cranberry juice

INTERVENTIONS:
Other: cranberry juice — 27% cranberry juice

SUMMARY:
This protocol is a clinical trial to validate proanthocyanidin A2 (PAC-A2) as a useful marker of cranberry intake. We hypothesize the consumption of this cranberry beverage in a progressive dosing schedule will increase PAC-A2 excretion in urine. Five generally healthy, nonsmoking, pre-menopausal women (absent major chronic diseases including cardiovascular, endocrine, gastrointestinal, and renal conditions), age 20-40 years, with a body mass index (BMI) of 18.5-25 kg/m2 will be recruited from the Boston area because sexually active women in this age range are particularly vulnerable to urinary tract infection. Volunteers will be asked to consume their assigned cranberry beverage at a dose of 8 oz/day according to a weekly dosing schedule. Relevant clinical information and eleven 24-hour and morning spot urine samples each will be collected from subjects during the study. Urinary PAC-A2 concentration will then be determined to validate if it can serve as a marker of compliance of cranberry juice consumption.

DETAILED DESCRIPTION:
People who frequently eat whole grains, fruits and berries, vegetables, beans and legumes, nuts, seeds, cocoa, tea, wine, and fruit or vegetable juices may have decreased risk of diseases. It is believed that some of these health benefits are due to phytochemicals present in these foods and beverages. Phytochemicals are nutrients that are naturally present in plant-based foods and beverages. Recently, cranberry containing foods and beverages are believed to prevent urinary tract infection. However, how cranberry decrease urinary tract infection is not very clear. To better understand how phytochemicals in cranberries may benefit health, we want to learn how they are absorbed and eliminated from the body. Thus, the purpose of the main study is to see whether we can measure phytochemicals from cranberries in health volunteers after they drink cranberry juice.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy premenopausal women
* aged 20-40 y
* body mass index (BMI): 18.5-25 kg/m2
* sexually active but not pregnant or planning to become pregnant
* no advance plans to discontinue use of hormonal contraceptives if they are taken

Exclusion Criteria:

* Use of medications known to affect lipid metabolism
* History of a bilateral mastectomy
* Use of medications known or suspected to influence blood pressure
* cardiovascular diseases
* Gastrointestinal diseases,
* Renal or chronic kidney disease
* Endocrine disorders
* Rheumatologic diseases
* Immune deficiency conditions
* Active treatment for cancer of any type longer than 1 y
* Systolic blood pressure >139 mmHg and/or diastolic blood pressure >89 mmHg
* Regular use (more than 1x/wk) of any acid-lowering medications, laxatives (including fiber supplements) or anti-diarrheal medications
* Use of any antibiotics in the last month
* Regular use of systemic steroids, oral or injectable
* Gain or loss of more than 5% of body weight in the last 6 mo
* Any history of or known allergies to cranberries or cranberry products
* Regular use of any dietary supplements containing vitamins, minerals, herbal or other plant-based preparations, fish oil supplements or homeopathic remedies.
* Usual daily ethanol intake of equal and more than 2 drinks
* Cigarette smoking and/or nicotine replacement use.
* Strict vegetarians (vegans)
* Pregnancy
* Infrequent (<3/wk) or excessive (>3/d) number of regular bowel movements
* Inability to discontinue or refrain from ASA/NSAID or Tylenol use for 72 h prior to and for the duration of testing on Visits 2-13
* Participation in a clinical research trial within 60 d of their enrollment visit (Visit 2)
* Specific laboratory blood or urine analysis parameters of: Creatinine >1.5 mg/dL, Electrolytes, calcium, phosphorous - out of normal ranges, ALT and AST >1.5 nmol, Total bilirubin - above normal range, Fasting glucose ≥126 mg/dL, Total cholesterol >239 mg/dL, Triglycerides ≥300 mg/dL, CBC: HCT <32% for females, below normal range for males, WBC, PLT - out of normal range, hematuria, proteinuria

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cranberry Juice
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cranberry Juice
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (3.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Proanthocyanidin A2
Description: proanthocyanidin A2 concentration in urine is determined using a LC-MS/MS method.
Time Frame: 24-hour urine and morning spot urine
Population: The subjects included 5 generally healthy premenopausal women, age 20-40 y, with a body mass index (BMI) ranging from 18.5 to 25 kg/m2. The specific operational criteria used to assess eligibility included: age, BMI, premenopausal status, not pregnant or planning to become pregnant.
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Cranberry Juice
Number analyzed (Participants) | 5
ng/mg creatinine
  24 h urine | 0.6 (0.5)
  morning spot urine | 0.20 (0.16)

ADVERSE EVENTS:
Time Frame: The whole intervention duration was 8 weeks.
Arm/Group | Cranberry Juice
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No